CLINICAL TRIAL: NCT03173807
Title: Prostate Nutrition and Exercise STudy (ProNEST)
Acronym: ProNEST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find adequate funding
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer McArdle, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCI 16-172
Record Dates: First submitted 2017-05-24; First posted 2017-06-02 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Metabolic Syndrome; Prostate Cancer; Diet Modification
MeSH Terms: conditions — Metabolic Syndrome; Prostatic Neoplasms | interventions — Diet

STUDY DESIGN:
Intervention Model Description: This is a pilot study that will employ a randomized, 2-arm wait-control design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary and exercise counseling (Active Comparator): The duration of study in Arm A will be 24 months, with study assessments and interventions (review of diet, food diary, and guidance from the dietician; review of activity journal, assessment of body composition, tests for gait, balance and muscle strength, and new assignment from the exercise trainer) done at baseline, 3 months, 6 months, 12 months and 24 months.
  Interventions: Behavioral: diet and exercise guidance and modifications
- standard of care (Active Comparator): The duration of study in Arm B will be 24 months, with study assessments and interventions (review of diet, food diary, and guidance from the dietician; review of activity journal, assessment of body composition, tests for gait, balance and muscle strength, and new assignment from the exercise trainer) done at baseline, 12 months, 15 months, 18 months and 24 months. At 12 months, participants in Arm B will be offered the same intervention that Arm A received during months 1-12.
  Interventions: Behavioral: diet and exercise guidance and modifications

INTERVENTIONS:
Behavioral: diet and exercise guidance and modifications — Review of diet, food diary, and guidance from the dietician; review of activity journal, assessment of body composition, tests for gait, balance and muscle strength, and new assignment from the exercise trainer

SUMMARY:
The purpose of this study is to test the feasibility of nutrition and exercise counseling program for reducing the incidence of metabolic syndrome in prostate cancer patients on Androgen Deprivation Therapy.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the role of dietary modifications and exercise in patients started on ADT for preventing and or delaying metabolic syndrome in this aging population. The study will employ a randomized, 2-arm wait-control design. Subjects will be randomized in a 1:1 ratio into two arms: dietary modifications and exercise counseling (Arm A) or standard of care (Arm B). The duration of intervention in Arm A will be 24 months. At 12 months, participants in Arm B will be offered the same intervention that Arm A received during months 1-12. Medical records will be accessed up to 5 years for standard of care visits. The goal of this project is to generate preliminary data on the feasibility of applying such an intervention on a much bigger population with approximately 100 subjects on each arm. For this pilot, we aim to randomize 20 patients to each arm. The principal investigator or co-investigators who are evaluating the patient will perform the randomization since this is an open-label, non-therapeutic study. The ADT received by patients on both arms is considered standard of care therapy for their prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written, informed consent
2. 18 years of age or greater
3. Histologically or biochemically confirmed hormone-naïve prostate adenocarcinoma
4. Recently started or re-started ADT within 4 months of starting the study
5. Eastern Oncology Co-operative Group (ECOG) performance 0-1
6. Patient who is on an antihypertensive medications with a blood pressure less than 130 systolic and 85 mm Hg diastolic
7. Patient who is on an antihyperlipidemic agents with TG ≤ 150 mg/dl, serum HDL ≥40 mg/dL

Exclusion Criteria:

1. Current use of taxane based chemotherapy for metastatic disease
2. Clinically significant or active cardiovascular disease:

   1. No previous MI within the past 12 months
   2. No uncontrolled angina within 12 months
   3. History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
   4. Uncontrolled hypertension (systolic BP > 170 mmHg or diastolic BP > 100 mmHg at screening)
   5. CHF with NYHA class 3 or 4
3. Structurally unstable bone lesions suggesting impending fracture
4. Estimated life expectancy of < 6 months
5. Patients who meet criteria for metabolic syndrome that are uncontrolled based on the Internal Diabetes Federation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The disease under study is prostate cancer
Enrollment: 0 (Actual)
Dates: Start 2017-08-31 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of metabolic syndrome in Arm A as compared to Arm B at 12 months | 12 months
  Metabolic syndrome will be defined by the following measurements: weight circumference, BMI, blood tests (Fasting glucose, Hemoglobin A1c, Lipid Panel, LDH and blood pressure), blood pressure. The information will be collected from medical records of standard of care visits

SECONDARY OUTCOMES:
Quality of life assessment | 24 months
  Quality of life assessed by the FACT-P (version 4) questionnaire
Patient activity | 24 months
  Patient activity using wearable tracking devices and questionnaire
Physical function and performance | 24 months
  Performance testing will be done using the following measure: short physical performance battery of balance, gait speed measuring physical function, and chair stand measuring lower body muscular endurance; an arm curl test measuring upper body muscular endurance, back scratch test measuring upper body flexibility, and chair sit-and-reach test measuring lower body flexibility. Anthropometric measurements will be completed measuring body mass index, abdominal girth with measuring tape.
Body composition | 24 months
  Body composition with a bioelectrical impedance analyzer. Body fat composition using skin calipers will also be measured
Adherence to treatment plan | 24 months
  Adherence to treatment plan by diet diary, pedometer and activity journal

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McArdle, PA-C, Principal Investigator — UPMC CancerCenter

IPD SHARING:
Plan to Share IPD: No